CLINICAL TRIAL: NCT04285463
Title: Defining Optimal Settings for Transbronchial Lung Cryobiopsy II: An Ex-Vivo Human Lungs Model Study for Improvement of Specimen Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Moishe Liberman, Thoracic Surgeon Principal Investigator, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19.280
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Transbronchial Lung Cryobiopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transbronchial Lung Cryobiopsy (TBLC) — TBLC is a relatively new endoscopic technique used to obtain lung parenchyma specimens. It is a minimally invasive technique performed with a flexible or rigid bronchoscope under deep sedation or general anesthesia. Flexible cryoprobes of either 1.9 or 2.4 mm in diameter are introduced into a bronchoscope and a compressed gas, most commonly carbon dioxide or nitrous oxide, is released at high flow at the tip of the probe. As the tissue rapidly freezes, it adheres to the probe and is avulsed and extracted with a quick pullback movement followed by immediate extraction of samples.

SUMMARY:
Diffuse parenchymal lung disease (DPLD) or Interstitial Lung Disease (ILD) comprises a broad variety of lung pathologies in which accurate diagnosis is crucial given to the different prognosis and therapeutic approaches, especially with the advent of new antifibrotic therapies.

Histology is an important tool when radiologic findings, clinical manifestations and bronchoalveolar lavage analysis are inconclusive. Surgical lung biopsy (SLB) is the gold standard for tissue sampling/analysis, however there is an associated cost and risk with a mortality-related between 1.8 and 3.6% for elective cases and up to 16% for the non-elective ones.

Transbronchial lung cryobiopsy (TBLC) is a safe, well-established technique used to obtain lung biopsies with large, high-quality specimens using compressed gas to freeze the tissue. The larger fragments do not contain the same crush artifacts seen in conventional transbronchial biopsies (TBB), but the non-standardization of the technique could be a limitation to the quality of the specimens and its safety.

The objective of this project is to determine the optimal settings for TBLC in human lungs with ILD in order to obtain the best quality specimens with the lowest risk profile. Two previous studies using animal models evaluated the technical components, such as probe size, freezing time and probe to pleura distance that results in good quality specimens. However, these were in normal animal lungs without ILD. In this new project, multiple TBLCs will be taken from lungs of documented ILD patients undergoing lung transplantation after their removal from the recipient patient at the time of lung transplantation.

DETAILED DESCRIPTION:
Transbronchial lung cryobiopsy (TBLC) is a less invasive procedure than surgical lung biopsy (SLB) to establish the diagnosis of interstitial lung disease (ILD) and as an endoscopic intervention can be done as an outpatient procedure. This technology has also being used for cryoadhesion to remove tissue from the airway. The freeze lung tissue provides bigger samples than the conventional transbronchial lung biopsy (TBB), less crush artifacts with more alveolar structures which gives better quality specimens and diagnostic yield for ILDs that usually has a complex morphologic pattern like unusual interstitial pneumonia and nonspecific interstitial pneumonia compared by TBB forceps biopsy. A recent trial showed that the histological diagnosis was obtained in only 34.1% of patients who had a TBB and the diagnostic yield of this technique was 29.1%. Lung cryobiopsy is associated with higher diagnostic yield (up to 83%) than TBBs and because of this, TBB is not recommended for ILD diagnosis in the current guidelines.

The diagnostic algorithm for ILD etiology definition is complex and has been born out of the necessity for diagnosis in patients where gold standard lung biopsy is associated with significant risk and therefore is typically saved as a last resort. Currently, SLB is indicated in only about 4 to 5% of the new cases suspected to have ILD. If TBLC is shown to be associated with lower complication rates, the investigator may be able to obtain definitive histological diagnoses in a great majority of cases and forego complex, inefficient and inaccurate methods of disease diagnosis. However, in order to replace SLB, TBLC should provide a similar diagnostic yield and better safety profile. Compared to SLB, retrospective data has shown that TBLC is associated with fewer complications, lower mortality, and better patient tolerance and recently one multicentric prospective trial (COLDICE) was designed to compare both techniques and guide the diagnostic accuracy for TBLC, not yet known. Several groups have published retrospective series of TBLC in ILD with promising results and diagnostic yields, however, the different technical components for performing a TBLC are very heterogeneous among the published series. Probe size, freezing time and distance from the probe to pleura are all parameters that may influence the size and quality of the samples.

As a technique recently applied to obtain adequate lung tissue for ILD differential diagnosis, its use was first described in 2009, there is no standard way to perform TBLC, and very limited data on how these parameters can influence biopsy quality. It is not clear which settings or parameters could affect the results. A few animal studies documented positive correlation between freezing time and biopsy size in TBLC. Published series on humans have used 4 and 6 seconds with a mini-cryoprobe probe and between 1 to 2 cm from the visceral pleura.

One of the limitations from the previous studies was that the lung specimens were obtained from healthy animal lungs. The lungs from patients undergoing transplant are affected by diffuse parenchymal pathologies and should offer a good predictor of how to obtain the best specimens for highest diagnostic yield in human lungs. The ex-vivo human model also has the advantage of performing multiple lung biopsies without any risks related with the procedure in in-vivo patients.

ELIGIBILITY:
Inclusion Criteria:

* Lungs from patients undergoing lung transplantation after their removal from the recipient patient with previous informed consent signed before transplantation.

Exclusion Criteria:

* Patients not candidates for surgical removal of the lungs during the act of transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Determine the probe size that yield the best lung biopsy specimens for histological analysis in an ex-vivo human model. | Time of procedure
  Multiple Transbronchial Lung Cryobiopsies (TBLCs) will be taken from the lungs using different probe sizes: 1.9 and 2.4 milimeters .
  The size and quality of the lung tissue samples will be compared to analyze which settings are optimal for obtaining the best quality specimens.
Determine the freezing probe time that yield the best lung biopsy specimens for histological analysis in an ex-vivo human model. | Time of procedure
  Multiple Transbronchial Lung Cryobiopsies (TBLCs) will be taken from the lungs and during the procedure each probe (1.9 and 2.4 milimiters) will be activated with different freezing times: first with 30 seconds followed by 20 seconds, then 10 seconds, 5 seconds and 3 seconds, successively.
  The size and quality of the lung tissue samples will be compared to analyze which settings are optimal for obtaining the best quality specimens.
Determine the distance from tip of the probe to the pleura that yield the best lung biopsy specimens for histological analysis in an ex-vivo human model. | Time of procedure
  Multiple Transbronchial Lung Cryobiopsies (TBLCs) will be taken from the lungs and during the procedure each probe (1.9 and 2.4 milimiters) will be activated at different distances from the pleura Inside the bronchus: first 5 milimeters apart, then 10 milimeters and 20 milimeters, successively.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quéebec, Canada

IPD SHARING:
Plan to Share IPD: No